CLINICAL TRIAL: NCT05862207
Title: Prevalence and Risk Factors of Nephrocalcinosis in Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mena Saad Mohamed, resident doctor, Sohag University
Other Study IDs: Nephrocalcinosis in children
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Nephrocalcinosis
MeSH Terms: conditions — Nephrocalcinosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study prevalence, risk factors, possible etiologies, clinical presentation and outcome of nephrocalcinosis in children at Sohag University Hospital.

DETAILED DESCRIPTION:
Nephrocalcinosis (NC) is characterized by deposition of calcium salts in the renal parenchyma. It is classified by ultrasonography into three types: cortical, medullary, and diffuse nephrocalcinosis . Cases of nephrocalcinosis in children are increasing and are becoming common causes for hospital admissions or visits to renal clinics. In addition, it is associated with significant long-term sequelae, including morbidity caused by recurrent stones as well as the development of chronic kidney disease (CKD).

The exact pathogenesis of nephrocalcinosis remains under investigation, in medullary nephrocalcinosis the main cause is hypercalciuria. Increased urinary calcium load arises either through increased calcium absorption (extra-renal causes) or impaired calcium reabsorption within the renal tubule . The majority of calcium reabsorption (~65%) occurs in the proximal tubule, and (~25%) is reabsorbed in the thick ascending limb of the loop of Henle and (~5%) is reabsorbed from the cortical collecting duct . Identification of monogenic causes of nephrocalcinosis affecting these areas has provided valuable insights into the pathogenesis of this heterogeneous condition. Interestingly, although a further (~7-10% (of calcium is reabsorbed within the distal convoluted tubule, no monogenic causes of nephrocalcinosis have been identified which affect this section of the renal Tubule . Nephrocalcinosis can occur due to various metabolic or renal tubular disorders, Vitamin D excess, medication, and prematurity .

The condition can progress to chronic kidney disease (CKD), and the renal prognosis is determined by its underlying cause, so a diagnostic evaluation in all children with NC to determine its causes and preserve kidney function is mandatory . Since the use of kidney ultrasound (US) as a routine diagnostic procedure, NC is detected in growing numbers of children. There is Different incidence rates and etiologies are reported in children with NC, reflecting the difference in geographic, genetic, and socioeconomic back ground.

Classifications of NC, based on its US appearance, have been proposed, distinguishing medullary, cortical and global NC . It has also been stated that whether NC is harmful or not depends on its magnitude, and on whether it is the result of an ongoing problem or of a transient insult .

Diagnosis of nephrocalcinosis is important to stop progression of renal injury. A detailed history should be obtained, including birth history, diet, fluid intake, medications, vitamin supplementation, developmental history, and other known diseases or conditions. A detailed family history also is very important. Physical examination findings are typically nonspecific, but the presence of signs that are syndromic in nature may provide helpful information to narrow the differential diagnosis .

ELIGIBILITY:
Inclusion Criteria:

* • All patients aged from one month to 12 years diagnosed with nephrocalcinosis at pediatric department and nephrology outpatient clinic.

Exclusion Criteria:

* • Children with nephrolithiasis without nephrocalcinosis.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all infants and children diagnosed with nephrocalcinosis and followed up at our pediatric nephrology clinic and pediatric department at Sohag University Hospitals during the study duration
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
percentage of nephrocalcinosis among renal diseases | one year
  percentage of children presented with nephrocalcinosis among all children with renal diseses in sohag university hospital

SECONDARY OUTCOMES:
Percentage of each risk factor of Nephrocalcinosis | one year
  percentage of each risk factor related to Nephrocalcinosis in children in ssohag univesity hospital

REFERENCES:
- [Result] Monet-Didailler C, Chateil JF, Allard L, Godron-Dubrasquet A, Harambat J. [Nephrocalcinosis in children]. Nephrol Ther. 2021 Feb;17(1):58-66. doi: 10.1016/j.nephro.2020.12.001. Epub 2021 Jan 15. French. PMID 33461896
- [Result] Hoppe B, Martin-Higueras C, Younsi N, Stein R. [Nephrolithiasis and nephrocalcinosis in children and adolescents]. Urologie. 2022 Oct;61(10):1099-1109. doi: 10.1007/s00120-022-01888-3. Epub 2022 Jul 8. German. PMID 35925106
- [Result] Habbig S, Beck BB, Hoppe B. Nephrocalcinosis and urolithiasis in children. Kidney Int. 2011 Dec;80(12):1278-91. doi: 10.1038/ki.2011.336. Epub 2011 Sep 28. PMID 21956187